CLINICAL TRIAL: NCT00385242
Title: PET and Recovery Following Revascularization: Outcome and Cost-effectiveness of FDG PET in Left Ventricular Dysfunction (PARR 2)
Brief Title: PET and Recovery Following Revascularization (PARR 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Rob Beanlands, Rob S. Beanlands, MD, FRCPC, Chief of Cardiology, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MCT-37412
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Coronary Artery Disease; Ventricular Dysfunction, Left
Keywords: coronary artery disease; left ventricular dysfunction; positron emission tomography; viable myocardium; revascularization; cost effectiveness
MeSH Terms: conditions — Coronary Artery Disease; Ventricular Dysfunction, Left | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PET guided Therapy (Active Comparator): Patients will be randomized to undergo positron emission tomography aspart of their clinical work up
  Interventions: Procedure: Positron emission tomography: FDG viability imaging; Other: PET imaging
- Standard care (Active Comparator): Patients will be randomized to standard care will under go other types of imaging or work up for revascularization without PET imaging.
  Interventions: Other: PET imaging

INTERVENTIONS:
Procedure: Positron emission tomography: FDG viability imaging — FDG PET viability imaging
  Arms: PET guided Therapy
Other: PET imaging — PET viability imaging

SUMMARY:
Rationale: Patients with severe ventricular dysfunction and coronary disease have high morbidity and mortality. They may benefit from revascularization, but have significant peri-operative morbidity and mortality. Positron emission tomography (PET) imaging with F-18-fluorodeoxyglucose (FDG) can detect viable myocardium that may recover from revascularization in such patients. It is unclear whether use of FDG PET in this population is improves outcome or is cost-effective.

Objectives: The principal aim is to determine whether FDG PET-guided therapy is effective versus standard care. Secondary objectives are to determine whether FDG PET-guided therapy improves LV function, quality of life and is good value for money versus standard care.

DETAILED DESCRIPTION:
Patients with severe ventricular dysfunction and coronary artery disease have high morbidity and mortality but may benefit from revascularization. However, there is also significant peri-operative morbidity and mortality among these patients. This accounts for the variable approach to these patients in different cardiac centres. Clearly this patient group has the most to gain when coronary revascularization is beneficial, but also the most to lose when it is not helpful. There is a need for an approach that can better define patients with severe ventricular dysfunction due to ischemia, who will be more likely to benefit from revascularization. Positron emission tomography (PET) imaging with F-18-Fluorodeoxyglucose (FDG) has been used to evaluate patients with ventricular dysfunction, to detect ischemic but viable myocardium more likely to recover from revascularization. Recently retrospective studies have shown that FDG PET can identify patients at high risk for cardiac events if they do not undergo revascularization. However, these studies did not evaluate whether FDG PET actually directed therapy decisions and because of their study design, could not determine whether FDG PET altered patient outcome. Our recent studies have shown that FDG PET can have important impact on therapy decisions and that patients with ischemic but viable myocardium are at increased risk. However it remains unclear whether an approach which utilizes FDG PET to define ischemic but viable myocardium can have a beneficial effect on patient outcome. It is also important to consider the potential clinical impact of FDG PET balanced against its limited availability. In addition, despite the cost of the technology, preliminary data from our group and others suggest a potential cost savings. Accordingly, a prospective randomized study is needed to evaluate whether FDG PET directed therapy has a beneficial effect on patient outcome and is cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years of age.
* Documented ejection fraction of <35% attributable to CAD.
* Documented CAD
* Any patient being considered for revascularization, transplant/heart failure work up or where, in the opinion of the attending physician or surgeon, viability imaging would be considered useful in ongoing clinical management decisions.

Exclusion Criteria:

* Other co-morbid conditions making survival unlikely
* < 6 weeks post myocardial infarction
* CAD unsuitable for revascularization
* emergency revascularization is required.
* severe valvular disease that requires surgery.
* Geographically inaccessible
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2000-06; Primary Completion 2006-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
time to occurence of the composite clinical endpoint of cardiac death,myocardial infarction, transplantation, or re-hospitalization for unstable angina or heart failure. | 5 years

SECONDARY OUTCOMES:
occurrence of the composite endpoint; individual components of the composite endpoint; quality of life, costs, and cost-effectiveness of PET-guided therapy versus control. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rob SB Beanlands, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Beanlands RS, Nichol G, Huszti E, Humen D, Racine N, Freeman M, Gulenchyn KY, Garrard L, deKemp R, Guo A, Ruddy TD, Benard F, Lamy A, Iwanochko RM; PARR-2 Investigators. F-18-fluorodeoxyglucose positron emission tomography imaging-assisted management of patients with severe left ventricular dysfunction and suspected coronary disease: a randomized, controlled trial (PARR-2). J Am Coll Cardiol. 2007 Nov 13;50(20):2002-12. doi: 10.1016/j.jacc.2007.09.006. Epub 2007 Oct 10. PMID 17996568
- [Background] D'Egidio G, Nichol G, Williams KA, Guo A, Garrard L, deKemp R, Ruddy TD, DaSilva J, Humen D, Gulenchyn KY, Freeman M, Racine N, Benard F, Hendry P, Beanlands RS; PARR-2 Investigators. Increasing benefit from revascularization is associated with increasing amounts of myocardial hibernation: a substudy of the PARR-2 trial. JACC Cardiovasc Imaging. 2009 Sep;2(9):1060-8. doi: 10.1016/j.jcmg.2009.02.017. PMID 19761983
- [Background] Abraham A, Nichol G, Williams KA, Guo A, deKemp RA, Garrard L, Davies RA, Duchesne L, Haddad H, Chow B, DaSilva J, Beanlands RS; PARR 2 Investigators. 18F-FDG PET imaging of myocardial viability in an experienced center with access to 18F-FDG and integration with clinical management teams: the Ottawa-FIVE substudy of the PARR 2 trial. J Nucl Med. 2010 Apr;51(4):567-74. doi: 10.2967/jnumed.109.065938. Epub 2010 Mar 17. PMID 20237039
- [Background] Shukla T, Nichol G, Wells G, deKemp RA, Davies RA, Haddad H, Duchesne L, Freeman M, Gulenchyn K, Racine N, Humen D, Benard F, Ruddy TD, Chow BJ, DaSilva J, Garrard L, Guo A, Chen L, Beanlands RS. Does FDG PET-assisted management of patients with left ventricular dysfunction improve quality of life? A substudy of the PARR-2 trial. Can J Cardiol. 2012 Jan-Feb;28(1):54-61. doi: 10.1016/j.cjca.2011.09.012. Epub 2011 Dec 3. PMID 22138342
- [Derived] Mc Ardle B, Shukla T, Nichol G, deKemp RA, Bernick J, Guo A, Lim SP, Davies RA, Haddad H, Duchesne L, Hendry P, Masters R, Ross H, Freeman M, Gulenchyn K, Racine N, Humen D, Benard F, Ruddy TD, Chow BJ, Mielniczuk L, DaSilva JN, Garrard L, Wells GA, Beanlands RS; PARR-2 Investigators. Long-Term Follow-Up of Outcomes With F-18-Fluorodeoxyglucose Positron Emission Tomography Imaging-Assisted Management of Patients With Severe Left Ventricular Dysfunction Secondary to Coronary Disease. Circ Cardiovasc Imaging. 2016 Sep;9(9):e004331. doi: 10.1161/CIRCIMAGING.115.004331. PMID 27609816